CLINICAL TRIAL: NCT01950286
Title: Four Years Experience With Hyper-CVAD Treatment of Adult T-cell Acute Lymphoblastic Leukemia in Sweden. Population-based Data.
Brief Title: Hyper-CVAD Treatment of Adult T-cell Acute Lymphoblastic Leukemia in Sweden.
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Piotr Kozlowski, MD, Region Örebro County
Other Study IDs: SVALL-02
Record Dates: First submitted 2013-09-07; First posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: T-cell Acute Lymphoblastic Leukemia
Keywords: T-cell Acute Lymphoblastic Leukemia; chemotherapy; allogeneic stem cell transplantation
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Hyper-CVAD (a chemotherapy regimen) has shown promising results in adult T-cell Acute Lymphoblastic Leukemia (T-ALL). Patients with T-ALL diagnosis were reported to the Swedish Adult Acute Leukemia Registry between October 2002 and September 2006. Hyper-CVAD was recommended to all patients without severe comorbidity. Allogeneic stem cell transplantation was recommended for patients with high-risk disease. The aim of this population-based study was to assess the efficacy of Hyper-CVAD treatment.

DETAILED DESCRIPTION:
Patients with T-ALL diagnosis were prospectively reported to the Swedish Adult Acute Leukemia Registry between October 2002 and September 2006. Missing data were complemented retrospectively. Hyper-CVAD (fractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone alternating with cycles of high-dose methotrexate and cytarabine) was recommended to all patients without severe comorbidity. Allogeneic stem cell transplantation (SCT) was recommended for patients with high-risk disease: white blood cell count >100×109/L, complete remission (CR) achievement after more than two courses, high minimal residual disease level, and relapsed disease (after CR2 achievement). In patients without high-risk factors maintenance therapy was given with per oral mercaptopurine and methotrexate for two years including reinduction courses: daunorubicine, vincristine and prednisolone every second month (1st year) and cytarabine, thioguanine and prednisolone every third month (2nd year).

ELIGIBILITY:
Inclusion Criteria: all patients with T-ALL diagnosis

Exclusion Criteria: no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T-ALL diagnosis reported to the Swedish Adult Acute Leukemia Registry between October 2002 and September 2006
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2002-10; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
overall survival | The outcome was assesed from T-ALL diagnosis to date of death or last follow-up (up to 125 months). Diagnosis was made between October 2002 and September 2006. All surviving patients were followed up until February 2013.
  Overall survival was defined as time from T-ALL diagnosis to the date of death from any cause or the date of last follow-up. All events (death/relapse) were reported prospectively to the the swedish acute leukemia registry.
  Inclusion Criteria: All patients with T-ALL diagnosis. Exclusion Criteria: No

SECONDARY OUTCOMES:
leukemia free survival | The outcome was assesed from T-ALL diagnosis to date of death or last follow-up (up to 125 months). Diagnosis was made between October 2002 and September 2006. All surviving patients were followed up until February 2013.
  Leukemia free survival was defined as time from achievement of complete remission to the date of T-ALL relapse or date of death from any cause or date of last follow-up. All events (death/relapse) were reported prospectively to the the swedish acute leukemia registry.
  Inclusion Criteria: All patients with T-ALL diagnosis. Exclusion Criteria: No

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kozlowski, MD, Principal Investigator — Orebro University Hospital, Orebro University
Locations (1):
- Orebro University Hospital, Örebro, Örebro County, Sweden